CLINICAL TRIAL: NCT03291808
Title: Pilot of Lifestyle and Asthma Intervention
Acronym: PLAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Lung Association (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Vermont (Other); University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00141509; R34HL136755 (NIH)
Record Dates: First submitted 2017-09-21; First posted 2017-09-25 (Actual); Results first posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-08

CONDITIONS: Asthma
Keywords: Obesity; Asthma; Weight loss
MeSH Terms: conditions — Asthma; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weight loss intervention (Experimental): Such designs are widely used in efficiently informing decisions to proceed to Phase III clinical trials. This trial design is appropriate when the effect of the placebo arm can reasonably be estimated (weight loss is likely to be close to 0), and the toxicity of the treatment is minimal (no toxicity is anticipated related to weight loss).18 Therefore, this will be a single arm 6-month study of 40 participants (20 at each site). All participants will be assigned to the weight loss intervention.
  Interventions: Behavioral: Weight loss intervention

INTERVENTIONS:
Behavioral: Weight loss intervention — This 6-month intervention will include restricted calorie intake and increased physical activity. Key behavioral strategies to facilitate changes in dietary habits and activity patterns will be introduced, promoted and reinforced throughout the program. Weekly "group meetings" in a synchronous chat (i.e., in real time) led by a facilitator will be the venue for the group process. Extensive web-based resources to support behavior changes will be offered. Group chat sessions will meet online weekly for 6 months.

SUMMARY:
This is to pilot test a weight loss intervention in obese patients with poorly controlled asthma.

Obesity is a risk factor for the development of asthma (approximately 250,000 cases per year of asthma in the U.S. are related to obesity).

Investigators' ultimate purpose is to test the hypothesis that weight loss through an intensive life style intervention will improve asthma control. But investigators first need to establish whether the weight loss intervention is effective in patients with asthma.

Objectives

1. The primary objective of this study is to determine the effectiveness of an internet-based weight loss intervention in producing weight loss in obese patients with poorly controlled asthma.
2. The ultimate purpose is to implement a multi-center weight loss intervention trial for obese patients with poorly controlled asthma.

DETAILED DESCRIPTION:
This will be a pilot study of a weight loss intervention at two centers, the University of Arizona and the University of Vermont. The primary outcome of interest will be the percent of participants achieving a 5% weight loss, which is the amount of weight loss that prior studies suggest is required to improve asthma control.

This will be a single arm-phase II futility trial; the "futility" to be assessed is the ability to produce weight loss. Such designs are widely used in efficiently informing decisions to proceed to Phase III clinical trials. This trial design is appropriate when the effect of the placebo arm can reasonably be estimated (weight loss is likely to be close to 0), and the toxicity of the treatment is minimal (no toxicity is anticipated related to weight loss). This is a 6-month study of 40 participants (20 at each site). All participants will be assigned to the weight loss intervention, which is described in detail below

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of asthma on regular prescribed controller therapy for at least 3 months
* Age: ≥18 years of age
* Obese: BMI > 30 kg/m2
* Poorly controlled asthma

  * Asthma Control Test Score < 19,19,20 or
  * Use of rescue inhaler, on average, > 2 uses/week for preceding month, or
  * Nocturnal asthma awakening, on average,1 or more times / week in preceding month, or
  * Emergency Department (ED)/hospital visit or prednisone course for asthma in past six months
* Ability and willingness to provide informed consent
* Ability to access internet weight loss program for trial period
* Completion of asthma diary cards and weight loss diary cards for same 3 consecutive days at visit 2

Exclusion Criteria:

* Prior history of bariatric surgery
* Any condition that puts the participant at risk from participation in a weight loss study or a condition that precludes participation in regular exercise as judged by the site physician.
* Pregnancy (by patient self-report)
* Participation in another weight loss intervention within the last month
* Weight loss of ≥ 10 pounds in the last 6 months by self-report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Dixon, MD, Principal Investigator — University of Vermont; Robert Wise, MD, Principal Investigator — Johns Hopkins School of Medicine; Janet Holbrook, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johnson O, Gerald LB, Harvey J, Roy G, Hazucha H, Large C, Burke A, McCormack M, Wise RA, Holbrook JT, Dixon AE. An Online Weight Loss Intervention for People With Obesity and Poorly Controlled Asthma. J Allergy Clin Immunol Pract. 2022 Jun;10(6):1577-1586.e3. doi: 10.1016/j.jaip.2022.02.040. Epub 2022 Mar 15. PMID 35304842
- See also: Related Info — http://medlineplus.gov/asthma.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-three were enrolled in the weight loss intervention in five cohorts, four English speaking and one Spanish speaking. Ten subjects dropped out before study completion, four reported this was related to research burden and six were lost to follow up: 33 participants completed the 6-month study. Recruitment was conducted at University of Vermont and University of Arizona.
Pre-assignment Details: Forty-eight participants were screened for the study intervention and entered a 4-week run-in period; five were excluded from enrolling into the weight loss intervention because they did not complete three consecutive days recording food intake, physical activity, weight and asthma symptoms.
Groups:
- Weight Loss Intervention: This trial design is appropriate when the effect of the placebo arm can reasonably be estimated (weight loss is likely to be close to 0), and the toxicity of the treatment is minimal (no toxicity is anticipated related to weight loss). Therefore, this will be a single arm 6-month study of 40 participants (20 at each site). All participants will be assigned to the weight loss intervention. Such designs are widely used in efficiently informing decisions to proceed to Phase III clinical trials.
  Weight loss intervention: This 6-month intervention will include restricted calorie intake and increased physical activity. Key behavioral strategies to facilitate changes in dietary habits and activity patterns will be introduced, promoted and reinforced throughout the program. Weekly "group meetings" in a synchronous chat (i.e., in real time) led by a facilitator will be the venue for the group process. Extensive web-based resources to support behavior changes will be offered. Group chat sessions will meet online weekly for 6 months.
Period: Overall Study
Arm/Group | Weight Loss Intervention
Started | 43
Completed | 33
Not Completed | 10
Not completed — Lost to Follow-up | 6
Not completed — Research burden | 4

BASELINE CHARACTERISTICS:
Population: People with poorly controlled asthma with a BMI of greater than 30
Arm/Group | Weight Loss Intervention
Number analyzed (Participants) | 43
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [41 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43
Forced Expiratory Vital Capacity % [Median (Inter-Quartile Range); unit: Percent predicted] | 80 [69 to 97]
Forced Vital Capacity % [Median (Inter-Quartile Range); unit: Percent predicted] | 85 [77 to 98]
Forced Expiratory Vital Capacity/Forced vital capacity [Median (Inter-Quartile Range); unit: Percent predicted] | 79 [71 to 83]
Asthma Control Test (ACT) [Median (Inter-Quartile Range); unit: units on a scale] — range 5-25, higher score indicative of better health
  units on a scale | 14 [12 to 17]
Asthma Symptom Utility Index, ASUI [Median (Inter-Quartile Range); unit: units on a scale] — range 0-1, higher score is indicative of better health
  units on a scale | .6 [.5 to .8]
Marks Asthma Quality of Life Questionnaire [Median (Inter-Quartile Range); unit: units on a scale] — Range, 1-80, lower score is indicative of better health
  units on a scale | 28 [18 to 41]
Standard Brief activity survey (SBAS) [Count of Participants; unit: Participants] — SBAS is used to categorize patients based on activity level into:
  * Inactive
  * Light Intensity
  * Moderate Intensity
  * Hard Intensity
  * Very Hard Intensity
  Participants
    Inactive | 11
    Light intensity | 23
    Moderate Intensity | 6
    Hard Intensity | 1
    Very Hard intensity | 1
    Unknown | 1
SF-36 Short forrm Survey Instrument [Median (Inter-Quartile Range); unit: units on a scale] — Range 0-100, higher score is indicative of better health
  units on a scale | 53 [43 to 68]
Impact of Weight on Quality of Life-Lite [Median (Inter-Quartile Range); unit: units on a scale] — Range 0-100, higher score is indicative of better health
  units on a scale | 55 [35 to 75]
Treatment Motivation and Readiness (TRE-MORE) [Median (Inter-Quartile Range); unit: units on a scale] — range 0-5, higher score is indicative of better health
  units on a scale | 3 [3 to 3]
Systemic corticosteroids [Count of Participants; unit: Participants]
  yes | 29
  no | 14

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss
Description: The primary outcome of interest will be the percent of participants achieving a 5% weight loss, which is the amount of weight loss that prior studies suggest is required to improve asthma control.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Weight Loss Intervention
Number analyzed (Participants) | 43
Participants | 43
Statistical Analysis 1: Comparison: Weight Loss Intervention; Test type: Other; p = .35, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Weight Loss Intervention
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 11/43
Other Adverse Events (participants affected / at risk) | 6/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Loss Intervention (N=43)
Asthma Exacerbations (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Emergency Department visit (General disorders) | 4 (11)
Small bowel obstruction (Gastrointestinal disorders) | 2 (3)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Chest pain with other symptoms (Cardiac disorders) | 1 (6)
Fall (General disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
(General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Loss Intervention (N=43)
Chest pain with other symptoms (General disorders) | 6 (6) — Other symptoms such as fall, hypertension, allergic reaction, knee pain, unknown

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT03291808/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT03291808/ICF_001.pdf